CLINICAL TRIAL: NCT04095117
Title: Evaluation of Sagittal Abdominal Diameter as a Predictor of the Skin to Epidural Space Distance in Obese Patients
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sameh M. Hakim, Professor of Anesthesiology, Intensive Care and Pain Management, Ain Shams University
Other Study IDs: FMASU MD 153/2019
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Epidural; Anesthesia, Headache
MeSH Terms: conditions — Obesity; Headache | interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Epidural block — Epidural catheter will be inserted at the L3-L4 or L4-L5 interspace in obese subjects scheduled for surgery on the lower extremities under epidural anesthesia.
  The sagittal abdominal diameter, BMI and skin to epidural space distance will be recorded.

SUMMARY:
The aim of this study is to evaluate the use of the sagittal abdominal diameter (SAD) as a potential predictor of the skin to epidural space distance (SESD) and to compare its accuracy versus that of the BMI as a previously validated predictor

DETAILED DESCRIPTION:
Adult patients from either sex with BMI from 30-39.9 kg/m², scheduled for lower abdominal operations or surgeries on the lower extremities under epidural anesthesia will be eligible. Pregnant women will be excluded.

The sagittal abdominal diameter (SAD), which is the anteroposterior diameter of the abdomen in the supine position at L4-5 level will be measured in all subjects along with the BMI prior to epidural placement.

The epidural space will be accessed at the L3-L4 or L4-L5 interspace with a 16-G or 18-G Tuohy needle using a loss of resistance to saline technique. The proper placement of the needle in the epidural space will be confirmed by connecting the hub of the epidural needle via a rigid extension tubing to a saline filled pressure transducer to demonstrate the characteristic epidural space pressure wave changes described by Arnuntasupakul and his colleagues (2016), which is a pulsatile waveform synchronized with arterial pulsations.

The distance from skin to epidural space will be marked on the needle with a sterile marker and will be recorded.

An epidural catheter will be passed into the epidural space and the epidural block will be activated in the usual way until adequate sensory and motor block is established in both lower extremities (Bromage score 3-4).

Successful placement of the epidural needle will be considered if the following two criteria are fulfilled: (1) Detection of the characteristic epidural pressure wave form as described above and (2) Establishment of adequate sensory and motor block.

Simple linear regression will be used to deduce an equation relating the skin to epidural space distance to the sagittal abdominal diameter or to the BMI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* BMI 30 to 39.9
* Either sex
* Elective surgery on lower extremities performed under epidural anesthesia

Exclusion Criteria:

* Pregnant women
* Contraindications to epidural block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects with BMI of 30 to 39.9 kg/m2 who are scheduled for lower extremity surgery under epidural anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the sagittal abdominal diameter for prediction of the skin to epidural space distance | 18 months
  Actual skin to epidural space distance will be determined and regressed on the sagittal abdominal diameter to determine accuracy of the latter for prediction of the former

SECONDARY OUTCOMES:
Accuracy of the BMI for prediction of the skin to epidural space distance | 18 months
  Actual skin to epidural space distance will be determined and regressed on the BMI to determine accuracy of the latter for prediction of the former

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided